CLINICAL TRIAL: NCT04680117
Title: Defining the Severe Paediatric Asthma Endotype: an Integrated Approach Combining Phenotypic Analyses Related to Immune, Metabolomics and Microbial Features
Brief Title: Defining the Severe Paediatric Asthma Endotype
Acronym: SevAsthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP200135; 2020-A00248-31 (Other: ID-RCB Number)
Record Dates: First submitted 2020-09-14; First posted 2020-12-22 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Severe Asthma
Keywords: Asthma; Severe; Immunologic; Metabolomic; Microbiologic profil
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases with SA, classified by age group (Other): Patient hospitalized for assessment of severe asthma
  Interventions: Other: Blood collection; Other: Saliva sample; Other: Nasal
- Controls among children w/ SA: frequent&infrequent exacerbators (Other): Frequent exacerbators have 2 or more asthma severe exacerbations in the past years
  Interventions: Other: Blood collection; Other: Saliva sample; Other: Nasal

INTERVENTIONS:
Other: Blood collection — Blood collection with samples of 15ml max by subject (case or control) at J0, M6 and M12:
  * subject less than 5 kg : 1.8 to 4.5 ml max
  * subject 5 kg to 10 kg : 4.5 to 9 ml max
  * subject 10 kg to 15 kg : 9 to 13.5 ml
  * subject 15 kg to 20 kg : 13.5 to 15 ml max
Other: Saliva sample — Saliva sample by subject at J0
Other: Nasal — Nasal brushing by subject at J0

SUMMARY:
The primary objective of this project is to extensively characterize the endotypes of pre-schoolers (0 to 6 years) and school-age children (6 to 12 years) with SA using an integrated approach, combining a description of their phenotype (asthma symptoms, atopy, and lung function) associated with histological (airway inflammation and remodelling), immune (innate and adaptive immunity), metabolomics, and microbiota analyses. This goal shall be achieved by an unsupervised in-depth analysis of patients requiring bronchial endoscopy, with bronchial alveolar lavage (BAL) and bronchial biopsy, as part of their clinical assessment.

DETAILED DESCRIPTION:
Asthma is a chronic disease affecting approximately 235 million people worldwide, and the number is rising. Asthma is not just a public health problem for developed countries; its incidence is also elevated in developing countries. Asthma concerns all age groups, but often starts in childhood. SA in children is infrequent, affecting 2-5% of the asthmatic paediatric population. Children with SA experience frequent SA attacks and have a reduced quality of life . They account for approximately half of the asthma healthcare costs. Asthma has long been thought to be a single disease but is now considered to encompass various conditions characterized by the same symptoms (wheeze, cough, shortness of breath, chest tightness), variable degrees of airflow limitation, and different pattern of inflammation. Recent studies highlighted the heterogeneity of asthma, and the potential influence of various pathogenic mechanisms, including airway inflammation, remodelling, and immune and metabolic pathways in a specific microbial environment. However, there is very little data concerning the pathological process, especially in children. Most of the data describing different asthma endotypes in children are derived from large observational prospective cohorts. Although very informative, these studies were designed to analyse a small number of easily measured parameters, mainly lung function and atopy. The complexity of asthma pathogenesis was therefore underestimated and the individuals' specificities only partially considered. In clinical practice, children with SA require an endoscopy, with broncho-alveolar lavage fluids (BALF) collection and bronchial biopsies to exclude a differential diagnosis and assess airway inflammation and remodelling. This approach also underestimates other components of the endotypes and results in "one size fits all" management based on high doses of inhaled steroids and the use of expensive biotherapy, such as anti-IgE therapy. Thus, although hospital admission and mortality ratesfor asthma decreased until the early 2000's, they have remained stable over the past 10 years. It is therefore imperative to develop new approaches that incorporate relevant parameters analysed in the airways. This project proposes an in-depth analysis, not only of clinical and functional parameters, but also of immune cells, metabolomic compounds, and microbiota present in the airways of asthmatic children.

The primary objective of the project is to extensively characterize the endotypes of pre-schoolers (0 to 6 years) and school-age children (6 to 12 years) with SA using an integrated approach, combining a description of their phenotype (asthma symptoms, atopy, and lung function) associated with histological (airway inflammation and remodelling), immune (innate and adaptive immunity), metabolomics, and microbiota analyses.

This goal shall be achieved by an unsupervised in-depth analysis of patients requiring bronchial endoscopy, with bronchial alveolar lavage (BAL) and bronchial biopsy, as part of their clinical assessment. The main hypothesis is that the complementarity of those approaches will allow investigators to delineate the immune and metabolic pathways and microbiota involved in children with SA. The secondary objectives are to: (1) cluster all data obtained to define new patient groups and develop biomarkers that summarise the different clusters; (2) determine the immune, metabolomic, and microbiota profile of these children to aid future fundamental research that will focus on dissecting new mechanisms involved in paediatric asthma; (3) determine whether pre-schoolers and school-age children with SA share common endotypic features; and (4) establish the basis for the prospective follow-up of patients to identify endotypes that predict asthma persistence throughout childhood, severity, and response to treatment.

ELIGIBILITY:
Patient Inclusion Criteria:

* Minors aged 0 to 6 years or 6 to 12 years, hospitalized for assessment of Severe Asthma
* Minors need with his follow-up an bronchial endoscopy with realization of LBA and biopsies of bronchial mucosa
* Social insurance affiliation, except AME
* Parents or legal guardians signed the Informed consent form

Control Inclusion Criteria:

* Minors aged 0 to 6 years or 6 to 12 years, hospitalized for assessment of severe respiratory syndrome except severe asthma
* Minors need with his follow-up an bronchial endoscopy with realization of LBA and biopsies of bronchial mucosa
* Social insurance affiliation, except AME
* Parents or legal guardians signed the Informed consent form

Patient Exclusion Criteria

* Prematurity (<37 weeks gestation)
* Broncho-pulmonary dysplasia, immune deficits, non-Severe Asthma bronchopathies, cystic fibrosis, heart disease, ongoing biotherapy

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Description of the environment and smoke exposure | 1 day
  Environment Living in a urban or non-urban area : n (%) Visible mold/dampness at home: n (%) Pet ownership: : n (%) Smoke exposure : n (%) Presence of pets at home : n (%)
Description of family atopy status | 1 day
  Atopy in 1 or 2 parents or siblings: n (%) Parental asthma : n (%) Parental atopic dermatitis: n (%) Parental immediate food allergy: n (%) Parental allergic rhinitis: n (%) Asthma in siblings: n (%) Atopic dermatitis in siblings: n (%) Immediate food allergy in siblings: n (%) Allergic rhinitis in siblings: n (%)
Description of Demographics | 1 day
  Sex male or female: n (%) Age at inclusion: y Weight (kg) Height (m) Body mass index : calculated from weight and height Atopy : n (%) Total IgE : n (%)
  * 1 positive allergy tests (SPT or sp IgE) to airborne allergens : n (%)
  * 1 positive SPT or sp IgE to food allergen: n (%) History of food allergy: n (%) History of allergic rhinitis: n (%) History of atopic dermatitis: n (%) Symptomatic gastro-oesophageal reflux: n (%)
Description of Asthma history in the past year | 1 day
  No of severe exacerbations : n
  ≥ 2 or 3 severe exacerbations: n (%) No. of cumulated days of oral steroids: n No. of emergency visits for acute asthma : n Asthma control ACT score : n
Description of Lung function | 1 day
  Lung function FEV1 pre-BD (% predicted) FEV1 post-BD (% predicted) FEV1 pre-BD (Zscore) FEV1 post-BD (Zscore) FEV1/FVC pre-BD (%) FEV1/FVC post-BD (%) FEV1/FVC pre-BD (Zscore) FEV1/FVC post-BD (Zscore) Post BD FEV1 reversibility (%) No of patients with reversibility : n (%) FeNO (ppb) Asthma therapy ICS : (%) ICS doses : µg/day. eq Budesonide ICS + LABA : n (%) Leukotriene modifier : n (%) Maintenance oral corticosteroids: n (%) Immunotherapy: n (%) Omalizumab or biologics: n (%)
Description of Asthma therapy | 1 day
  ICS : (%) ICS doses : µg/day. eq Budesonide ICS + LABA : n (%) Leukotriene modifier : n (%) Maintenance oral corticosteroids: n (%) Immunotherapy: n (%) Omalizumab or biologics: n (%)
Description of Airway remodeling | 1 day
  reticular basement membrane thickness expressed in µm; airway smooth muscle area ; epithelial integrity; vessel number; mucus gland area
Description of inflammatory and histological features in bronchoalveolar lavages (BAL) | 1 day
  Number of eosinophils, neutrophils, macrophages, basophils, lymphocytes expressed as percentage of total cells in BAL
Description of inflammatory and histological features in bronchial mucosa | 1 day
  Number of eosinophils, neutrophils, macrophages, basophils, lymphocytes expressed per square millimeters of submucosal area
Bronchial mucosa analysis | 1 day
  The number of IgE stained with anti-IgE Ab in the submucosa and the epithelium will be assessed and expressed per square millimeters of submucosal area The expression of cytokines in the mucosa will be assessed by multiplex and expressed in pg/ml or ng/ml.
  Quantify by quantitative PCR mRNA encoding cytokines, chemokines and others immune activation markers as relative mRNA levels.
BAL analysis | 1 day
  The number of mast cells, lymphocytes, innate lymphoid cells, mucosalassosiated invariant T (MAIT) cells, gammadelta T cells expressed as percentage of total cells in BAL, concentrations of Immunoglobulins G, E, M will be assessed and express in Ku/L The expression of cytokines will be assessed by multiplex and expressed in pg/ml or ng/ml.
Blood analysis | 1 day
  Number of eosinophils, neutrophils, macrophages, basophils, lymphocytes, innate lymphoid cells expressed as percentage of total cells in blood; number of mucosal associated invariant T (MAIT) cells will be assessed and expressed as percentage of total cells and T cells in blood The number of invariant natural killer T cells will be assessed and expressed as percentage of total cells and T cells in blood The number of gammadelta T cells will be assessed and expressed as percentage of total cells and T cells in blood The concentrations of Immunoglobulins G, E, M will be assessed and express in Ku/L The expression of cytokines will be assessed by multiplex and expressed in pg/ml or ng/ml.
Metabolomic signature | 1 day
  The global concentration of metabolites is first expressed as the signal intensity compared to internal controls. When metabolites are identified, they are quantified and their concentration expressed as pg/ml.
Microbiota analysis | 1 day
  Quantify by quantitative PCR mRNA and DNA encoding as relative mRNA and DNA levels

SECONDARY OUTCOMES:
Cluster analysis | 1 year
  Identify the main phenotypes of severe asthma by the cluster analysis.
Number of severe exacerbations in the 12 months following the inclusion | 1 year
  Patients will be then categorized in frequent exacerbators and non-frequent exacerbators (n) according to their number of severe exacerbations in the 12 months following inclusion
Asthma Control Test (ACT) score 12 months after inclusion | 1 year
  from 0 to 27 (for children 4-11 years); from 5-25 for children 12 years and older - higher score is better control
Asthma control 12 months after inclusion | 1 year
  according to international guidelines : not controlled, partially controlled, controlled
Description of lung function 12 months after the inclusion | 1 year
  FEV1 pre-BD (% predicted); FEV1 post-BD (% predicted); FEV1 pre-BD (Zscore); FEV1 post-BD (Zscore); FEV1/FVC pre-BD (%); FEV1/FVC post-BD (%); FEV1/FVC pre-BD (Zscore); FEV1/FVC post-BD (Zscore); Post BD FEV1 reversibility (%); No of patients with reversibility : n (%); FeNO (ppb)
Number of severe exacerbations during the 1 year follow up | 1 year
Number of emergency department visits for acute asthma during the 1 year follow up | 1 year
Number of cumulated days of oral steroids for asthma exacerbations during the 1 year follow up | 1 year
Number of hospital admissions for acute asthma during the 1 year follow up | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lezmi, Doctor (PHU), Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Name: Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No